CLINICAL TRIAL: NCT00968682
Title: Detection of Cardiac Dysfunction in Patients Treated With Trastuzumab for HER-2 Positive Breast Cancer. The CADY Study
Brief Title: CADY Study ICORG 08-01
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: 08-01 ICORG; ICORG-08-01; EU-20948
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer; Cardiac Toxicity
Keywords: cardiac toxicity; HER2-positive breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Biological: trastuzumab
Other: laboratory biomarker analysis
Procedure: assessment of therapy complications

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with cancer treated with trastuzumab may help doctors learn more about biomarkers related to heart dysfunction. It may also help doctors predict which patients will develop heart dysfunction.

PURPOSE: This clinical trial is studying biomarkers to see how well they predict heart dysfunction in women with breast cancer treated with trastuzumab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To prospectively evaluate whether an increase in cardiac biomarker levels can predict cardiac dysfunction in women with HER2/neu-positive breast cancer treated with trastuzumab as curative intent.

Secondary

* To develop a predictive model for use in this patient population based on the most accurate and sensitive combination of biomarkers.

This is an observational study with all patients having

* Blood tests for BNP, Nt-pro BNP, CRP and Troponin-T every 42 days (6 weeks) whilst on treatment with chemotherapy and/or Trastuzumab.
* Echocardiograph or MUGA before treatment, after completion of anthracycline therapy where applicable, and every twelve weeks whilst on Trastuzumab. Assessment of ejection fraction may be carried out at any time for symptoms. All Echocardiographs and MUGAs will be carried out locally. 2-D Echocardiograph is the preferred method for assessment of LVEF. Where possible, the same cardiac imaging facility should be used for all LVEF assessments. A sample study from each participating institution will be reviewed by the principal investigating cardiologist. Results of left ventricular function assessment will be used to make treatment decisions as normal. Managing clinicians will not be made aware of the results of biomarker assessments, thus this study is blinded.
* Cardiorespiratory symptom assessment, ECOG score, vitals, weight and NYHA (if applicable) prior to each dose of anthracyclines and every 6 weeks whilst on Paclitaxel-trastuzumab and on single agent Trastuzumab.

Patients on BETH :

The LVEF monitoring sequence required by CADY will be altered to parallel that required by BETH. Thus, echocardiograph or MUGA will be carried out according to the BETH cardiac safety monitoring protocol. This altered schedule applies only to patients enrolled in both studies. Of note, for patients on the BETH study, all LVEF assessments must be performed by the same method used at baseline.

Patients on ALTTO:

It is possible that a patient who is enrolled on both CADY and ALLTO may not eventually receive Trastuzumab. Nonetheless, as Lapatinib is also associated with a risk of cardiotoxicity, such patients should remain on study whilst receiving single agent Lapatinib. The schedule of on study assessments will be identical to that of patients receiving Trastuzumab.

For patients enrolled in both studies, the LVEF monitoring sequence required by CADY will be altered to parallel that required by ALLTO. Thus, echocardiograph or MUGA will be carried out according to the ALLTO cardiac safety monitoring protocol Of note, for patients on the ALLTO study, all LVEF assessments must be performed by the same method used at baseline.

ELIGIBILITY:
Inclusion Criteria

1. HER-2 positive breast cancer by immunohistochemistry and/or fluorescence in-situ hybridisation.
2. Planned neoadjuvant and/or adjuvant treatment with chemotherapy and Trastuzumab either sequentially or in combination or single agent Trastuzumab.
3. 18 years of age or older.
4. Disease Stage I-III, whose treatment plan includes Trastuzumab either sequentially, in combination or as a single agent will be eligible for inclusion in the study.
5. As this is a non-interventional study, patients enrolled in therapeutic clinical trials will also be eligible for inclusion.
6. Treatment with curative intent.
7. ECOG Performance status 0, 1 or 2.
8. Adequate cardiac function, with MUGA or Echocardiograph > 50%.
9. Written informed consent.

Exclusion Criteria:

1. Presence of a medical or psychiatric condition, which, in the opinion of the investigator, would potentially pose a risk to the patient by participating in this trial.
2. Evidence of metastatic disease.
3. Patients with uncontrolled hypertension (sustained systolic blood pressure >180mmHg or diastolic blood pressure >100mmHg), significant valvular disease (aortic or mitral regurgitation of 3 or 4+/ 4+ severity or stenosis of either valve), history of uncontrolled cardiac arrhythmias, prior symptomatic or asymptomatic myocardial infarction or angina pectoris requiring anti-anginal medication.
4. Prior anthracycline or Trastuzumab therapy.
5. Inability to give informed consent for any reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HER2 positive breast cancer, who are foreseen for neoadjuvant and/or adjuvant treatment with chemotherapy and Trastuzumab either sequentially or in combination or single agent Trastuzumab.
  Patients enrolled on BETH or ALTTO are also eligible.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2008-04; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cardiac biomarker levels in predicting cardiac dysfunction | End of trial
Development of a predictive model for use based on the most accurate and sensitive combination of biomarkers | End of trial

CONTACTS AND LOCATIONS:
Overall Officials: Ray McDermott, MD, Principal Investigator — Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital
Locations (14):
- Ireland (14):
  - Bons Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Our Ladies of Lourdes Hospital, Drogheda
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Mater Private Hospital, Dublin
  - University College Hospital, Galway
  - Letterkenny General Hospital, Letterkenny
  - Mid- Western Regional Hospital, Limerick
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford